CLINICAL TRIAL: NCT00067808
Title: Phase II Randomized Study of Three Different Schedules of Low-Dose Decitabine (5-AZA-2'-Deoxycytidine) in Myelodysplastic Syndrome (MDS)
Brief Title: Study of Three Different Schedules of Low-Dose Decitabine in Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID03-0180
Record Dates: First submitted 2003-08-27; First posted 2003-08-28 (Estimated); Results first posted 2011-05-26 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia
Keywords: Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia; MDS; Decitabine; Dacogen; Methylation
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Decitabine 10 mg/m^2 IV (Active Comparator): 10 mg/m^2 intravenous (IV) over 1 hour daily for 10 days
  Interventions: Drug: Decitabine
- Decitabine 20 mg/m2 IV (Active Comparator): 20 mg/m2 IV over 1 hour daily for 5 days
  Interventions: Drug: Decitabine
- Decitabine 20 mg/m2 SQ (Active Comparator): 20 mg/m2 subcutaneous (SQ) daily for 5 days
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — 10 mg/m^2 by vein over 1 hour daily for 10 days
  Other Names: Dacogen
  Arms: Decitabine 10 mg/m^2 IV
Drug: Decitabine — 20 mg/m2 by vein (IV) over 1 hour daily x 5 days
  Other Names: Dacogen
  Arms: Decitabine 20 mg/m2 IV
Drug: Decitabine — 20 mg/m2 subcutaneous (SQ) daily x 5 days
  Other Names: Dacogen
  Arms: Decitabine 20 mg/m2 SQ

SUMMARY:
The goal of this clinical research study is to learn if decitabine (given at 3 different doses) can help to control Myelodysplastic Syndrome (MDS). The safety of these 3 treatments will also be studied.

DETAILED DESCRIPTION:
Treatment: Methylation is a change that occurs to Deoxyribonucleic acid (DNA) that has an effect on gene usage in human cells. Abnormal methylation is very common in leukemias. Decitabine is a new drug that blocks DNA methylation.

Before treatment starts, a physical exam, blood tests (between 4-6 tablespoons), and a bone marrow study will be done. To collect a bone marrow sample, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow is withdrawn through a large needle. Women able to have children must have a negative blood or urine pregnancy test.

When this study began, participants were randomly assigned (as in the toss of a coin) to one of 3 treatment groups. The assignment to one of the 3 schedules was adjusted according to how well patients respond to treatment. About 17 patients were assigned to each group for the first 50 patients.

Participants in the first group received decitabine intravenously (IV--through a needle in their vein) over one hour, once a day, for 10 days. Treatment was given every 4 to 8 weeks depending on how well their blood counts recovered. Participants in the second group received decitabine as an IV infusion over one hour, once a day, for 5 days. Treatment was given every 4 to 8 weeks. Participants who received decitabine by vein got the same total dose per course. Participants in the third group received decitabine by subcutaneous (SQ) injections (injections given under the skin) twice a day for 5 days. As in the first and second group, treatment was given every 4 to 8 weeks.

After 65 patients were enrolled on this study, it was decided that the 5-day IV schedule was the best of the 3 schedules. The study will now continue with all new patients receiving the 5 -day IV decitabine treatment. If you are now enrolling on the study, you will be placed in this treatment group, instead of being randomly assigned to a treatment group.

Participants who are already on study and who are receiving the 5-day SQ schedule or the 10-day IV schedule, will be given the option to change to the 5-day IV schedule at the start of their next course of study drug treatment, since this is considered the new "standard" schedule on this particular study.

If you choose to take part in this study and begin receiving the study treatment described above, your response to treatment will be checked after completing 8 weeks of therapy. If the response to treatment is good, treatment with decitabine will continue. Decitabine treatment may be continued for up to 24 courses, or as long as it is judged best to control the leukemia.

During this study, you will need to visit your doctor for a physical exam and vital signs. The frequency of doctor visits will vary depending on your physical condition, but will be required at least once a month.

Blood tests (about 2 teaspoons) will be done about every week during the first 6-8 weeks of treatment, then every 1 to 2 weeks for the length of the study. The blood samples will be used for routine lab tests. Periodic bone marrow samples will also be taken to check cells related to the disease before, during, and after completion of this study.

Patients will be taken off study if the disease gets worse or intolerable side effects occur.

This is an investigational study. Decitabine is not yet Food and Drug Administration (FDA) approved.Up to 133 participants will be treated in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. MDS and 5% or more marrow blasts, or IPSS risk intermediate 1-2 or high risk; or chronic myelomonocytic leukemia
2. Performance status 0-2 (Eastern Cooperative Oncology Group (ECOG) scale); adequate hepatic (bilirubin < 2 mg/dl) and renal functions (creatinine <2mg/dl); New York Heart Association (NYHA) cardiac status III-IV excluded.
3. Signed informed consent
4. No prior intensive combination chemotherapy or high-dose ara-C (>/= 1g/m2 per dose). Prior biologic therapies, targeted therapies and single agent chemotherapy allowed.
5. Patients must have been off chemotherapy for 2 weeks prior to entering this study and recovered from the toxic effects of that therapy, unless there is evidence of rapidly progressive disease. Use of Hydroxyurea for patients with rapidly proliferative disease is allowed for the first two weeks on therapy.

Exclusion Criteria:

1. Nursing and pregnant females are excluded. Patients of childbearing potential should practice effective methods of contraception. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
2. Patients with active and uncontrolled infections
3. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2003-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hagop M Kantarjian, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Oki Y, Jelinek J, Shen L, Kantarjian HM, Issa JP. Induction of hypomethylation and molecular response after decitabine therapy in patients with chronic myelomonocytic leukemia. Blood. 2008 Feb 15;111(4):2382-4. doi: 10.1182/blood-2007-07-103960. Epub 2007 Nov 30. PMID 18055864
- See also: M.D. Anderson Cancer Center's website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period 6/4/03 - 5/18/09; all patients were registered at The University of Texas M.D. Anderson Cancer Center.
Pre-assignment Details: Enrollment of 128 patients: 1 patient withdrew consent prior to treatment; 3 did not meet eligibility requirement for a total of 124 evaluable patients.
Groups:
- Decitabine 10 mg/m2 IV: 10 mg/m2 by vein (IV) over 1 hour daily for 10 days
Period: Overall Study
Arm/Group | Decitabine 10 mg/m2 IV | Decitabine 20 mg/m2 IV | Decitabine 20 mg/m2 SQ
Started | 17 | 93 | 14
Completed | 17 | 93 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decitabine 10 mg/m2 IV | Decitabine 20 mg/m2 IV | Decitabine 20 mg/m2 SQ | Total
Number analyzed (Participants) | 17 | 93 | 14 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 45 | 7 | 59
  >=65 years | 10 | 48 | 7 | 65
Age Continuous [Median (Full Range); unit: years] | 67 [44 to 90] | 65 [37 to 83] | 64 [51 to 79] | 65 [37 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 33 | 4 | 40
  Male | 14 | 60 | 10 | 84
Region of Enrollment [Number; unit: participants]
  United States | 17 | 93 | 14 | 124

OUTCOME MEASURES:

1. Primary Outcome: Participant Responses
Description: Objective responses by International Working Group criteria: 'Complete Response' (CR) defined as Normalization of the peripheral blood and bone marrow with <5% bone marrow blasts, a peripheral blood granulocyte count > (1.0 x 109/ L, and a platelet count > 100 x 109/L); 'Other Response' including Partial Remission (PR) defined as above, except for the presence of 6-15% marrow blasts, or 50% reduction if <15% at start of treatment combined with participants who meet all criteria for CR except for platelet recovery to >100 x 109/L; and 'No Response'.
Time Frame: Response to treatment after 8 weeks of therapy
Population: As treated: 124 patients completed treatment.
Measure: Number; unit: Participants
Arm/Group | Decitabine 10 mg/m2 IV | Decitabine 20 mg/m2 IV | Decitabine 20 mg/m2 SQ
Number analyzed (Participants) | 17 | 93 | 14
Participants
  Complete Response | 4 | 47 | 4
  Other Response | 6 | 21 | 4
  No Response | 7 | 25 | 6

ADVERSE EVENTS:
Time Frame: 6 Years
Arm/Group | Decitabine 10 mg/m2 IV | Decitabine 20 mg/m2 IV | Decitabine 20 mg/m2 SQ
Serious Adverse Events (participants affected / at risk) | 5/17 | 32/93 | 7/14
Other Adverse Events (participants affected / at risk) | 4/17 | 32/93 | 8/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine 10 mg/m2 IV (N=17) | Decitabine 20 mg/m2 IV (N=93) | Decitabine 20 mg/m2 SQ (N=14)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Adrenal Insufficiency (General disorders) | 0 (0) | 0 (0) | 1 (1)
Allergic Reaction (General disorders) | 0 (0) | 2 (2) | 0 (0)
Cardiac arrythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac Ischemia (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Cardipulmonary arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 6 (6) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Elevated cardiac triponin (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Encephalopathy (General disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Knee effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 4 (5) | 13 (17) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Prolonged myelosuppression (General disorders) | 0 (0) | 0 (0) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Supraventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (General disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine 10 mg/m2 IV (N=17) | Decitabine 20 mg/m2 IV (N=93) | Decitabine 20 mg/m2 SQ (N=14)
Allergic reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Elevated alanine aminotransferase (Hepatobiliary disorders) | 1 (1) | 9 (9) | 0 (0)
Anorexia (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0)
Elevated aspartate aminotransferase (Hepatobiliary disorders) | 1 (1) | 7 (7) | 0 (0)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1) | 8 (8) | 1 (1)
Elevated Creatinine (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 5 (5) | 1 (1)
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Mucositis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 12 (13) | 1 (1)
Pain (General disorders) | 0 (0) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No